CLINICAL TRIAL: NCT04624750
Title: An Open-label, Non-Comparative Study to Evaluate the Steady-State Pharmacokinetics, Safety, and Efficacy of Mexiletine in Adolescents and Children With Myotonic Disorders
Brief Title: Open Label Study in Adolescents and Children With Myotonic Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEX-NM-301
Record Dates: First submitted 2020-10-20; First posted 2020-11-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Mexiletine

STUDY DESIGN:
Intervention Model Description: This is an open-label, multi-centre, single arm, interventional, study to evaluate the safety, steady-state PK, and efficacy of mexiletine for the treatment of myotonia in paediatric population aged 6 to < 18 years.
  The study comprises a screening period of 30 days, a dose-titration period of 4 weeks, and a maintenance period of 4 weeks. After last visit, all patients will be offered follow-up in clinical study MEX-NM-303 (PIP Study 7).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 and 2 (Other): 7 patients aged 12 to < 18 years , inclusive in cohort-1 7 patients aged 6 to < 12 years, inclusive in cohort-2
  Interventions: Drug: Mexiletine

INTERVENTIONS:
Drug: Mexiletine — Patients will be enrolled sequentially into 2 cohorts. Cohort 1 - (patients aged 12 to < 18 years): approximately 8 weeks - 4 weeks of dose titration period + 4 weeks of maintenance period.
  Cohort 2 - (patients aged 6 to < 12 years,): approximately 8 weeks - 4 weeks of dose titration period + 4 weeks of maintenance period.
  Enrolment for Cohort 2 will begin after initial safety assessment of patients in Cohort 1 by the DSMB and no safety concerns are observed. The dose level for cohort 2 will be confirmed by PK modelling study.
  Other Names: Namuscla ™

SUMMARY:
This is an open-label, multi-centre, single arm, interventional study to describe the steady-state PK, safety, and efficacy of mexiletine in paediatric patients (6 to <18 years of age) with myotonic disorders.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, single arm, interventional study to describe the steady-state PK, safety, and efficacy of mexiletine in paediatric patients (6 to <18 years of age) with myotonic disorders.

Patients who meet the eligibility criteria will be enrolled stepwise, sequentially in 2 cohorts by age groups.

Cohort 1 - Adolescents aged 12 to <18 years, will be enrolled first. If no safety concerns are observed (based on data evaluation by the Data Safety Monitoring Board [DSMB]), and the dose for the age group 6 to <12 years is confirmed by PK model, enrolment for Cohort 2 will begin.

Cohort 2 - Children aged 6 to <12 years, will be enrolled. The overall treatment duration for each cohort will be approximately 56 days (8 weeks): a dose titration phase of 4 weeks and the maintenance phase of 4 weeks. The overall study duration would be approximately 22 months.

Dose titration phase: In this phase, patients will receive mexiletine starting at an age appropriate dose (as evaluated by the investigator and based on body weight) at a frequency of once a day. Dose will be up-titrated every 14 days based on tolerability of mexiletine up to a maximum of three-times a day as assessed by investigator.

Maintenance phase: During the maintenance phase, patients will continue to receive mexiletine at the best-tolerated dose from the titration phase for further 4 weeks. Following completion, all participants will be offered follow-up in PIP Study 7 (MEX-NM-303) (EudraCT: 2019-003758-97).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 6 and < 18 years who are able to comply with the study requirements
2. A genetically confirmed diagnosis of NDM or DM (DM1or DM2)
3. Presence of clinical symptoms of myotonia (hand grip myotonia, myotonia in the leg muscles, any other myotonia symptoms)
4. No significant cardiac abnormalities as determined by a cardiologist's assessment of the ECG and echocardiogram performed within 3 months prior to enrolment in the study. (If not done within 3 months before trial, electrocardiogram (ECG) and echocardiogram assessments will be performed at screening)
5. No history of any significant liver disorder
6. Patients receiving mexiletine treatment agree to stop treatment at least 7 days prior to initiation of treatment with Namuscla
7. Patients receiving other antimyotonic treatment agree to stop treatment for at least 7 times the half-life of respective drug
8. Laboratory investigations for haematology, biochemistry, and urinalysis at screening are within the normal range, or showing no clinically relevant abnormal values, as judged by the Investigator.
9. Female patients of childbearing potential must be using an acceptable form of birth control as determined by the Investigator (e.g., oral contraception, implantable, injectable/transdermal hormonal contraception, intrauterine device (IUD), barrier methods), tubal ligation or are practicing abstinence.
10. Patients able to provide assent to study participation and a parent or legal guardian to sign the written informed consent prior to study entry.

Exclusion Criteria:

1. Any contra-indication to mexiletine as listed in the Namuscla Summary of Product Characteristics (SmPC):

   1. Hypersensitivity to the active substance, or to any of the excipients
   2. Hypersensitivity to any local anaesthetic
   3. Ventricular tachyarrhythmia
   4. Complete heart block (i.e., third-degree atrioventricular block) or any heart block susceptible to evolve to complete heart block (first-degree atrioventricular block with markedly prolonged PR interval (≥ 200 ms) and/or wide QRS complex (≥ 120 ms), second-degree atrioventricular block, bundle branch block, bifascicular and trifascicular block),
   5. QT interval > 450ms
   6. Myocardial infarction (acute or past), or abnormal Q-waves
   7. Symptomatic coronary artery disease
   8. Heart failure with ejection fraction <50%
   9. Atrial tachyarrhythmia, fibrillation or flutter
   10. Sinus node dysfunction (including sinus rate < 50 bpm)

       • Co-administration with medicinal products inducing torsades de pointes (class Ia, Ic, III antiarrhythmics): Co-administration of mexiletine and antiarrhythmics inducing torsades de pointesclass Ia: quinidine, procainamide, disopyramide, ajmaline; class Ic: encainide, flecainide, propafenone, moricizine; class III: amiodarone, sotalol, ibutilide, dofetilide, dronedarone, vernakalant) increases the risk of potentially lethal torsades de pointes.
   11. Co-administration with medicinal products with narrow therapeutic index
2. Any other neurological or psychiatric condition that might affect the study assessments
3. Any clinically significant illness, laboratory findings, ECG, or other clinical symptoms, which in the opinion of the Investigator could affect the patient's optimal participation in the study
4. Strong inducer or inhibitor of CYP2D6 or CYP1A2 within 7 days prior to study drug administration
5. Any concurrent illness, or medications which could affect the muscle function
6. Seizure disorder, diabetes mellitus requiring treatment by insulin
7. Pregnant or breastfeeding
8. Concurrent participation in any other clinical trial.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Number and frequency of adverse events (AEs)/serious adverse events (SAEs) | Baseline to Day 56
  Number and frequency of adverse events (AEs)/serious adverse events (SAEs), throughout the study while on treatment with Namuscla
Incidence of adverse events of special interest (AESI) | Baseline to Day 56
  Incidence of adverse events of special interest (AESI)
Changes in ECG assessments from baseline | Baseline to Day 56
  On resting ECG any alteration will be noted:
  * Mild ECG abnormalities: PR interval ≥200 ms and QRS duration ≥100 ms
  * Severe ECG abnormalities: PR interval ≥240 ms, QRS duration ≥120 ms, second or third degree AV block and a rhythm other than sinus
Efficacy of Namuscla treatment on the clinical outcomes based on the following functional evaluation mean change in Visual Analogue Scale (VAS) for muscle stiffness. | Baseline to Day 56
  Mean change in Visual Analogue Scale (VAS) for muscle stiffness. The VAS is constructed as an absolute measure, with a 10 cm straight horizontal line having the endpoints "no stiffness at all" and "stiffness as worst possible". The patient's responses will be scored on the line to the nearest millimetre (a 100-point scale). (myotonia severity).
Efficacy of Namuscla treatment on the clinical outcomes(change from baseline to Days 14, 28, 42 and 56, respectively) based on the following functional evaluation | Baseline to Day 56
  The score of handgrip myotonia as quantitatively measured using a commercially available grip dynamometer and computerised capture system. In standardised conditions (i.e. in a room at controlled temperature, after a definite period of rest), maximum voluntary contractions following forced right hand grip will be recorded and the time to relax from 90% to 5% of maximal force will be determined using automated analysis software

SECONDARY OUTCOMES:
Mean change in VAS score for muscle pain, weakness and fatigue | Baseline - Day 56
  The VAS is constructed as an absolute measure, with a 10 cm straight horizontal line having the endpoints "no stiffness at all" and "stiffness as worst possible". The patient's responses will be scored on the line to the nearest millimetre (a 100-point scale). The score of stiffness severity as self-reported by the patient on a 10-point VAS will be used for adolescents and children older than 8 years and will be summarised descriptively by visit
Clinical myotonia assessment for mean change in time to open the eyes | Baseline - Day 56
  Mean change in time to open the eyes after forced eye closure as measured on a stopwatch (when eyelid myotonia present). Subjects will be asked to squeeze their eyes closed for 5 seconds then rapidly open them for 5 seconds then rapidly open. Five trials of each manoeuvre will be performed in sequence at each visit and the time measured on a stopwatch
Clinical myotonia assessment of clinical change in flexor myotonia | Baseline - Day 56
  Clinical change in flexor myotonia (right hand flexor muscles). Subjects will be asked to make a tight fist for 5 seconds then rapidly open. Five trials of each manoeuvre will be performed in sequence at each visit and the time measured on a stopwatch
Clinical myotonia assessment of mean change in time to perform Timed-up and go (TUG) test | Baseline - Day 56
  Mean change in time to perform Timed-up and go (TUG) test. Measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
Mean change in health-related quality-of-life as measured by the Paediatric Quality of Life (PedsQL) score | Baseline - Day 56
  Mean change from baseline to Day 56, respectively in health-related quality-of-life as measured by the Paediatric Quality of Life (PedsQL) score. These multidimensional scales assess the frequency of health problems using generic and disease-specific approaches, respectively. Subjects and/or parent or proxies report a score of 0 to 4 (never to almost always) and questionnaires are tailored to age groups.
Clinical Global Impression (CGI) scores (efficacy and tolerability) evaluated by the patient | Baseline - Day 56
  Clinical Global Impression (CGI) scores (efficacy and tolerability) evaluated by the patient, a parent or proxy and by the investigator at baseline and Day 56. Evaluated on a 4-point scale as very efficient, good, fair or poor.
Mean change in Myotonia Behaviour Scale (MBS) scores | Baseline - Day 56
  Mean change from baseline to Day 56 in Myotonia Behaviour Scale (MBS) scores The Myotonia Behaviour Scale (MBS) (Hammaren et al., 2005) 0 No stiffness
  1. Some stiffness exists, which can be ignored
  2. Some stiffness exists, which can be ignored at times, but doesn't impair daily activities
  3. Stiffness exists, which demands a higher level of mental awareness when performing some duties and activities
  4. Severe stiffness exists, which impairs every duty and activity
  5. Incapacitating stiffness exists, which demands constant moving not to be totally locked up, with regard to movement
Changes in clinical laboratory values for laboratory safety assessments - Potassium | Baseline - Day 56
  Changes in Potassium values from baseline to Day 56.
Acceptability of the capsule formulation with respect to the swallowability. | Baseline - Day 56
  Acceptability of the capsule formulation with respect to the swallowability. It will be assessed by interviewing patients and their caregivers at Day 56.
Palatability of alternative administration | Baseline - Day 56
  Palatability of alternative administration (capsule content with milk/juice or sprinkled on food) by 5-point facial hedonic scale correlated with 100-point Visual Analogue Scale (VAS) at each clinic visit
Changes in clinical laboratory values from baseline to Day 56 for laboratory safety assessments - Changes in Magnesium values | Baseline - Day 56
  Changes in Magnesium values from baseline to Day 56.
Changes in clinical laboratory values from baseline to Day 56 for laboratory safety assessments - Changes in Sodium values | Baseline - Day 56
  Changes in Sodium values from baseline to Day 56.
Changes in clinical laboratory values from baseline to Day 56 for laboratory safety assessments - Changes in Calcium values | Baseline - Day 56
  Changes in Calcium values from baseline to Day 56.
Changes in clinical laboratory values from baseline to Day 56 for laboratory safety assessments - Changes in Chloride values | Baseline - Day 56
  Changes in Chloride values from baseline to Day 56.
Mean change in Faces scale for muscle pain, weakness and fatigue | Baseline - Day 56
  A Faces (or other symbol) scale for children aged 6 to 8 years will be used to measure the score of muscle stiffness (myotonia severity). Faces scale will be used to assess pain, weakness and tiredness in study participants with a 10 cm straight horizontal line having the endpoints "no [symptom] at all" and "[symptom] as worst possible"

CONTACTS AND LOCATIONS:
Overall Officials: Christine Barnérias, MD, Principal Investigator — Hopital universitaire Necker-Enfants Malades
Locations (1):
- Hôpital Necker-Enfants-Malades, Paris, France